CLINICAL TRIAL: NCT04153773
Title: Retinal Thickness as a Potential Biomarker of Neurodegeneration and Early Cognitive Impairment in Patients With Multiple Sclerosis
Brief Title: OCT and Early Cognitive Impairment in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Esmael, Assistant Prof of Neurology, Mansoura University Hospital
Other Study IDs: Mansoura University Hospital 2
Record Dates: First submitted 2019-11-02; First posted 2019-11-06 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: 60 Patient
  Interventions: Diagnostic Test: OCT
- Group 2: 30 Control subject
  Interventions: Diagnostic Test: OCT

INTERVENTIONS:
Diagnostic Test: OCT — The degree of physical disability was assessed by using the Expanded Disability Status Scale (EDSS). The EDSS score ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
  Neurocognitive functions were evaluated using the Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS) that includes the following tests:
  1. Symbol Digit Modalities Test (SDMT) that is used for assessment of information processing speed.
  2. California Verbal Learning Test - 2nd edition (CVLT-II) .
  3. Brief Visuospatial Memory Test-Revised (BVMT-R)
  OCT assessment was performed by spectral domain-optical coherence tomography to assess the retinal nerve fiber layer thickness and macular volume in humans .
  Each eye for every patient was assessed by measuring the thickness of RNFL and GCC, respecting presence or absence of the previous history of optic neuritis (ON).
  Other Names: EDSS; Cognitive assessment

SUMMARY:
The aim of this study is to investigate the relationship between cognitive impairment and retinal nerve fiber layer & ganglion cell inner plexiform layer in MS.

DETAILED DESCRIPTION:
Cross-sectional study design, including 60 patients and 30 healthy controls. Subjects were investigated clinically, underwent retinal optical coherence tomography (OCT) and comprehensive cognitive assessments. The correlation between these modalities was evaluated by Spearman correlation.

ELIGIBILITY:
Inclusion Criteria:

* 60 MS patients diagnosed according to the revised McDonald criteria 2010 were included
* 30 healthy subjects with age and sex match control group.

Exclusion Criteria:

* Medical disorder other than MS that may grossly affect cognitive functions
* Pregnancy,
* Previous neurological or neuropsychiatric disorders,
* Alcohol or drug abuse,
* MRI findings which could not be attributed to MS.
* Severe visual disorders (> ± 6.0 dpt.)
* History of ocular surgery, glaucoma or diabetes.

Ages: 20 Years to 45 Years | Sex: All
Age Groups: Adult
Study Population: This was a cross-sectional study that was conducted in the Neurology Department of Mansoura University Faculty of Medicine, Egypt. 60 patients with MS were recruited from the period of Aug 2018 to September 2019.
  Participants 60 MS patients diagnosed according to the revised McDonald criteria 2010 were included . Both sexes aged 20-45 year were included.
  Age and sex matched the healthy control (HC) group which consisted of 30 subjects without any neurological or psychiatric disease and who were not related (within the first or second degree of consanguinity) to a patient with MS.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Optical coherence tomography | 24-48 hours
  OCT imaging was performed by spectral domain-optical coherence tomography to assess the retinal thickness.

SECONDARY OUTCOMES:
Cognitive assessment | 24-48 hours
  Neurocognitive functions were evaluated using the Brief International Cognitive Assessment for Multiple Sclerosis (BICAMS)
Expanded Disability Status Scale (EDSS) | 24 hours
  The EDSS score ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Esmael M Ahmed, MD, Principal Investigator — Assistant Prof of Neurology
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balk LJ, Sonder JM, Strijbis EM, Twisk JW, Killestein J, Uitdehaag BM, Polman CH, Petzold A. The physiological variation of the retinal nerve fiber layer thickness and macular volume in humans as assessed by spectral domain-optical coherence tomography. Invest Ophthalmol Vis Sci. 2012 Mar 9;53(3):1251-7. doi: 10.1167/iovs.11-8209. PMID 22266522
- [Result] Filippi M, Bar-Or A, Piehl F, Preziosa P, Solari A, Vukusic S, Rocca MA. Multiple sclerosis. Nat Rev Dis Primers. 2018 Nov 8;4(1):43. doi: 10.1038/s41572-018-0041-4. PMID 30410033
- [Result] Kalb R, Beier M, Benedict RH, Charvet L, Costello K, Feinstein A, Gingold J, Goverover Y, Halper J, Harris C, Kostich L, Krupp L, Lathi E, LaRocca N, Thrower B, DeLuca J. Recommendations for cognitive screening and management in multiple sclerosis care. Mult Scler. 2018 Nov;24(13):1665-1680. doi: 10.1177/1352458518803785. Epub 2018 Oct 10. PMID 30303036
- [Result] Rocca MA, Amato MP, De Stefano N, Enzinger C, Geurts JJ, Penner IK, Rovira A, Sumowski JF, Valsasina P, Filippi M; MAGNIMS Study Group. Clinical and imaging assessment of cognitive dysfunction in multiple sclerosis. Lancet Neurol. 2015 Mar;14(3):302-17. doi: 10.1016/S1474-4422(14)70250-9. Epub 2015 Feb 4. PMID 25662900
- [Result] Rocca MA, Battaglini M, Benedict RH, De Stefano N, Geurts JJ, Henry RG, Horsfield MA, Jenkinson M, Pagani E, Filippi M. Brain MRI atrophy quantification in MS: From methods to clinical application. Neurology. 2017 Jan 24;88(4):403-413. doi: 10.1212/WNL.0000000000003542. Epub 2016 Dec 16. PMID 27986875
- [Result] Kappos L, De Stefano N, Freedman MS, Cree BA, Radue EW, Sprenger T, Sormani MP, Smith T, Haring DA, Piani Meier D, Tomic D. Inclusion of brain volume loss in a revised measure of 'no evidence of disease activity' (NEDA-4) in relapsing-remitting multiple sclerosis. Mult Scler. 2016 Sep;22(10):1297-305. doi: 10.1177/1352458515616701. Epub 2015 Nov 19. PMID 26585439
- [Result] Perez Del Palomar A, Cegonino J, Montolio A, Orduna E, Vilades E, Sebastian B, Pablo LE, Garcia-Martin E. Swept source optical coherence tomography to early detect multiple sclerosis disease. The use of machine learning techniques. PLoS One. 2019 May 6;14(5):e0216410. doi: 10.1371/journal.pone.0216410. eCollection 2019. PMID 31059539
- [Result] Martinez-Lapiscina EH, Arnow S, Wilson JA, Saidha S, Preiningerova JL, Oberwahrenbrock T, Brandt AU, Pablo LE, Guerrieri S, Gonzalez I, Outteryck O, Mueller AK, Albrecht P, Chan W, Lukas S, Balk LJ, Fraser C, Frederiksen JL, Resto J, Frohman T, Cordano C, Zubizarreta I, Andorra M, Sanchez-Dalmau B, Saiz A, Bermel R, Klistorner A, Petzold A, Schippling S, Costello F, Aktas O, Vermersch P, Oreja-Guevara C, Comi G, Leocani L, Garcia-Martin E, Paul F, Havrdova E, Frohman E, Balcer LJ, Green AJ, Calabresi PA, Villoslada P; IMSVISUAL consortium. Retinal thickness measured with optical coherence tomography and risk of disability worsening in multiple sclerosis: a cohort study. Lancet Neurol. 2016 May;15(6):574-84. doi: 10.1016/S1474-4422(16)00068-5. Epub 2016 Mar 18. PMID 27011339
- [Result] London A, Benhar I, Schwartz M. The retina as a window to the brain-from eye research to CNS disorders. Nat Rev Neurol. 2013 Jan;9(1):44-53. doi: 10.1038/nrneurol.2012.227. Epub 2012 Nov 20. PMID 23165340
- [Result] Satue M, Obis J, Rodrigo MJ, Otin S, Fuertes MI, Vilades E, Gracia H, Ara JR, Alarcia R, Polo V, Larrosa JM, Pablo LE, Garcia-Martin E. Optical Coherence Tomography as a Biomarker for Diagnosis, Progression, and Prognosis of Neurodegenerative Diseases. J Ophthalmol. 2016;2016:8503859. doi: 10.1155/2016/8503859. Epub 2016 Oct 20. PMID 27840739
- [Result] Petzold A, Balcer LJ, Calabresi PA, Costello F, Frohman TC, Frohman EM, Martinez-Lapiscina EH, Green AJ, Kardon R, Outteryck O, Paul F, Schippling S, Vermersch P, Villoslada P, Balk LJ; ERN-EYE IMSVISUAL. Retinal layer segmentation in multiple sclerosis: a systematic review and meta-analysis. Lancet Neurol. 2017 Oct;16(10):797-812. doi: 10.1016/S1474-4422(17)30278-8. Epub 2017 Sep 12. PMID 28920886
- [Result] Serbecic N, Aboul-Enein F, Beutelspacher SC, Vass C, Kristoferitsch W, Lassmann H, Reitner A, Schmidt-Erfurth U. High resolution spectral domain optical coherence tomography (SD-OCT) in multiple sclerosis: the first follow up study over two years. PLoS One. 2011;6(5):e19843. doi: 10.1371/journal.pone.0019843. Epub 2011 May 17. PMID 21611198
- [Result] Balk LJ, Cruz-Herranz A, Albrecht P, Arnow S, Gelfand JM, Tewarie P, Killestein J, Uitdehaag BM, Petzold A, Green AJ. Timing of retinal neuronal and axonal loss in MS: a longitudinal OCT study. J Neurol. 2016 Jul;263(7):1323-31. doi: 10.1007/s00415-016-8127-y. Epub 2016 May 3. PMID 27142714
- [Result] Cruz-Herranz A, Balk LJ, Oberwahrenbrock T, Saidha S, Martinez-Lapiscina EH, Lagreze WA, Schuman JS, Villoslada P, Calabresi P, Balcer L, Petzold A, Green AJ, Paul F, Brandt AU, Albrecht P; IMSVISUAL consortium. The APOSTEL recommendations for reporting quantitative optical coherence tomography studies. Neurology. 2016 Jun 14;86(24):2303-9. doi: 10.1212/WNL.0000000000002774. Epub 2016 May 25. PMID 27225223
- [Result] Mendez-Gomez JL, Pelletier A, Rougier MB, Korobelnik JF, Schweitzer C, Delyfer MN, Catheline G, Monferme S, Dartigues JF, Delcourt C, Helmer C. Association of Retinal Nerve Fiber Layer Thickness With Brain Alterations in the Visual and Limbic Networks in Elderly Adults Without Dementia. JAMA Netw Open. 2018 Nov 2;1(7):e184406. doi: 10.1001/jamanetworkopen.2018.4406. PMID 30646353
- [Result] Cabrera DeBuc D, Gaca-Wysocka M, Grzybowski A, Kanclerz P. Identification of Retinal Biomarkers in Alzheimer's Disease Using Optical Coherence Tomography: Recent Insights, Challenges, and Opportunities. J Clin Med. 2019 Jul 9;8(7):996. doi: 10.3390/jcm8070996. PMID 31323964
- [Result] Polman CH, Reingold SC, Banwell B, Clanet M, Cohen JA, Filippi M, Fujihara K, Havrdova E, Hutchinson M, Kappos L, Lublin FD, Montalban X, O'Connor P, Sandberg-Wollheim M, Thompson AJ, Waubant E, Weinshenker B, Wolinsky JS. Diagnostic criteria for multiple sclerosis: 2010 revisions to the McDonald criteria. Ann Neurol. 2011 Feb;69(2):292-302. doi: 10.1002/ana.22366. PMID 21387374
- [Result] Kurtzke JF. Rating neurologic impairment in multiple sclerosis: an expanded disability status scale (EDSS). Neurology. 1983 Nov;33(11):1444-52. doi: 10.1212/wnl.33.11.1444. PMID 6685237
- [Result] Smith A. Symbol digit modalities test: manual. Western Psychological Corporation. Los Angeles (CA): Western Psychological Services; 2002.
- [Result] Delis DC, Kramer JH, Kaplan E, et al. California verbal learning test - second edition. Adult version. Manual. San Antonio (TX): The Psychological Corporation; 2000.
- [Result] Benedict RHB. Brief visuospatial memory testrevised. Odessa (Fla): Psychological Assessment Resources; 1997.